CLINICAL TRIAL: NCT06276452
Title: Supporting Resilience Among Re-entered Seniors
Acronym: SRRS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Louisville (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Stephanie Prost, Associate Professor, University of Louisville
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 23.0434; U2CDA050097 (NIH)
Record Dates: First submitted 2024-02-16; First posted 2024-02-26 (Actual); Last update posted 2025-03-26 (Actual); Status verified 2025-03

CONDITIONS: Chronic Disease
MeSH Terms: conditions — Chronic Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Supporting resilience psychoeducational group (Experimental): This group-based psychoeducational intervention will take place once weekly for eight weeks and will be centered upon building older adults' knowledge, skills, and motivation to manage chronic disease.
  Interventions: Behavioral: Psychoeducation

INTERVENTIONS:
Behavioral: Psychoeducation — Psychoeducation is the therapeutic management of illness through the increase of related knowledge, skills, and motivation.

SUMMARY:
The first goal (Aim 1) of this clinical trial is to learn about specific strengths, challenges, and desired areas of knowledge and skill-building among older adults who re-entered their communities from a period of incarceration and to then develop a new psychoeducational intervention tailored to these older adults. The second goal (Aim 2) of this clinical trial is to test if the intervention increases chronic disease management and whether the intervention is considered appropriate and acceptable by older adults who re-entered their communities from a period of incarceration.

Aim 1 participants will:

* complete a baseline survey
* participate in a focus group

Aim 2 participants will:

* complete a baseline survey
* participate in an 8-week once weekly intervention
* complete three follow up surveys

DETAILED DESCRIPTION:
The protocol for Aim 2 will be developed once the focus group data is analyzed.

ELIGIBILITY:
Inclusion Criteria:

* at least 45 years old
* have re-entered the community from a period of incarceration from jail or prison
* have at least one chronic health condition
* able to speak and understand English

Exclusion Criteria:

* aged 44 or younger
* have not re-entered the community from a period of incarceration from jail or prison
* does not have at least one chronic health condition
* unable to speak and understand English

Min Age: 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 8 (Estimated)
Dates: Start 2024-03-09 (Actual); Primary Completion 2026-11-30 (Estimated); Study Completion 2026-11-30 (Estimated)

PRIMARY OUTCOMES:
Chronic disease self managment | 12 weeks
  Patient-Reported Outcomes Measurement Information System (PROMIS) Self-Efficacy for Managing Chronic Conditions measures (viz. daily activities, medications and treatments, symptoms, emotions, social interactions)

CONTACTS AND LOCATIONS:
Locations (1):
- New Legacy Reentry, Louisville, Kentucky, United States

IPD SHARING:
Plan to Share IPD: No